CLINICAL TRIAL: NCT05089565
Title: Assessment of the Immune Response to SARS-CoV-2/COVID-19 Vaccination in Patients With Sarcoidosis
Brief Title: Immune Response to SARS-CoV-2/COVID-19 Vaccination in Sarcoidosis
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Foundation for Sarcoidosis Research (Other)
Responsible Party: Principal Investigator, Peter Sporn, MD, Professor of Medicine, Northwestern University
Other Study IDs: SP0069572
Record Dates: First submitted 2021-10-19; First posted 2021-10-22 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Sarcoidosis; SARS-CoV2 Infection; Vaccine Response Impaired
Keywords: sarcoidosis; SARS-CoV-2; vaccination; spike antibody; cell-mediated immune response; COVID-19; interferon-gamma
MeSH Terms: conditions — Sarcoidosis; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Serum, plasma, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sarcoidosis, not on treatment: Sarcoidosis patients, 18 years of age or older, not currently being treated with immunosuppressive medications
  Interventions: Diagnostic Test: Assay of (1) the level of anti-spike IgG antibody, and (2) interferon-gamma release in response to SARS-CoV-2 antigen stimulation
- Sarcoidosis, on treatment: Sarcoidosis patients, 18 years of age or older, currently being treated with immunosuppressive medications
  Interventions: Diagnostic Test: Assay of (1) the level of anti-spike IgG antibody, and (2) interferon-gamma release in response to SARS-CoV-2 antigen stimulation
- Healthy controls: Healthy individuals, matched for age and sex with those in the two sarcoidosis cohorts
  Interventions: Diagnostic Test: Assay of (1) the level of anti-spike IgG antibody, and (2) interferon-gamma release in response to SARS-CoV-2 antigen stimulation

INTERVENTIONS:
Diagnostic Test: Assay of (1) the level of anti-spike IgG antibody, and (2) interferon-gamma release in response to SARS-CoV-2 antigen stimulation — Measurement of humeral and cell-mediated immune responses to SARS-CoV-2 vaccination

SUMMARY:
People with sarcoidosis, particularly those with significant lung and/or cardiac involvement, who become infected with severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) are likely at increased risk of complications or death from COVID-19. While SARS-CoV-2 vaccines are highly efficacious in preventing COVID-19 in the general population, whether vaccination provides similar protection in people with sarcoidosis is unknown. The investigators hypothesize that people with sarcoidosis develop less robust antibody and cell-mediated immune responses to SARS-CoV-2 vaccination than healthy individuals, both as a consequence of the disease itself and due to treatment with immunosuppressive medications. This hypothesis will be examined by determining levels of anti-SARS-CoV-2 spike protein immunoglobulin G (IgG) antibody (Specific Aim 1) and measuring SARS-CoV-2-specific activation of peripheral blood T cells (Specific Aim 2) following SARS-CoV-2 vaccination in individuals with sarcoidosis treated and not treated with immunosuppressive medications, in comparison to age- and sex-matched healthy controls. For Specific Aim 1, a second-generation anti-SARS-CoV-2 spike IgG assay calibrated against an independent virus neutralization assay will be utilized. The results of this investigation will address a critical gap in the understanding of vaccine responses in people with sarcoidosis. In addition, the study will contribute knowledge needed to inform clinicians' recommendations to sarcoidosis patients regarding risk of infection after SARS-CoV-2 vaccination, and will help lay the basis for future trials to evaluate the possible benefit of vaccine boosters in individuals with poor immune responses to initial vaccination.

DETAILED DESCRIPTION:
Introduction, Hypothesis and Specific Aims

People with sarcoidosis, particularly those with significant lung and/or cardiac involvement, who become infected with SARS-CoV-2 are likely at increased risk of complications or death from COVID-19. While SARS-CoV-2 vaccines are highly efficacious in preventing COVID-19 in the general population, whether vaccination provides similar protection in people with sarcoidosis is unknown. The investigators hypothesize that people with sarcoidosis develop less robust antibody and cluster of differentiation 4 (CD4)+ T cell-mediated immune responses to SARS-CoV-2 vaccination than healthy individuals, both as a consequence of the disease itself and as a result of treatment with immunosuppressive medications.

Specific Aim 1. Determine blood anti-SARS-CoV-2 spike protein IgG antibody levels following SARS-CoV-2 vaccination in individuals with sarcoidosis treated and not treated with immunosuppressive medications, in comparison to age- and sex-matched healthy controls.

Specific Aim 2. Determine levels of SARS-CoV-2-specific activation of peripheral blood CD4+ T cells following SARS-CoV-2 vaccination in individuals with sarcoidosis treated and not treated with immunosuppressive medications, in comparison to age- and sex-matched healthy controls.

The results of this investigation will address a critical gap in the understanding of vaccine responses in people with sarcoidosis. In addition, the study will contribute knowledge needed to inform clinicians' recommendations to sarcoidosis patients regarding risk of infection after SARS-CoV-2 vaccination, and will help lay the basis for future trials to evaluate the possible benefit of vaccine boosters in individuals with poor immune responses to initial vaccination.

Background

The development of safe and effective vaccines against SARS-CoV-2 over the past year represents a scientific triumph and public health breakthrough in the battle to control the COVID-19 pandemic. Ongoing vaccination of the U.S. population has coincided with a >12-fold reduction in reported COVID-19 cases from a peak average of 260,000 per day in January 2021 to 21,000 per day as of this writing (May 29, 2021). Unfortunately, this has not been the case in other parts of the world, particularly low and middle income countries of the Global South, where vaccine availability has been severely limited and vaccination rates are so far quite low. Although less than the inequality internationally, there are disparities in vaccine access and uptake among groups within the U.S., with lower vaccination rates among African Americans, Latin Americans and others. As a result, members of these groups remain at increased risk, and will continue to sustain a disproportionate burden of COVID-19.

Another group at increased risk of developing COVID-19 is comprised of people with medical conditions or on treatments that cause immune suppression, who therefore may fail to mount a protective immune response to SARS-CoV-2 vaccination. For example, recent reports indicate that antibody responses to SARS-CoV-2 messenger RNA (mRNA) vaccines are suboptimal in substantial proportions of solid organ transplant recipients and patients with hematologic malignancies. Data on patients with connective tissue and other chronic inflammatory diseases are mixed, with some recent studies showing robust antibody responses to SARS-CoV-2 vaccines, even in those on immunosuppressive therapies, while another report found that antibody responses in such individuals are reduced and/or delayed. Notably, in the latter study, reduced antibody responses were associated the presence of an immune-mediated inflammatory disease, but not more likely in those on specific immunosuppressive medications. In contrast, another recent study found that use of methotrexate was associated with decreased antibody and cluster of differentiation 8 (CD8)+ T cell responses to the SARS-CoV-2 BNT162b2 mRNA vaccine, while other oral immunomodulatory drugs and tumor necrosis factor (TNF) inhibitors did not appear to have such an effect.

Whether the immune response to SARS-CoV-2 vaccination is impaired in people with sarcoidosis is not known. This is a critical question because sarcoidosis patients may be at increased risk for severe adverse outcomes of COVID-19. The literature on responses to other vaccines in sarcoidosis is sparse. One study reported no difference in the antibody response to influenza vaccination in untreated sarcoidosis patients compared to healthy controls. By contrast, in another report, antibody responses to tetanus vaccination were reduced in patients with sarcoidosis, 52% of whom were on oral corticosteroids, although the impairment in vaccine response was unrelated to corticosteroid therapy. There are no published data on T lymphocyte responses to vaccination in sarcoidosis, although the observation that CD4+ T cell activation and proliferation are impaired in active sarcoidosis suggests that the T cell response to SARS-CoV-2 vaccination may be reduced as well. In the absence of better data specific to the disease, a group of international experts recently put forward a strong recommendation for SARS-CoV-2 vaccination in people with sarcoidosis, and extrapolating from information on responses to other vaccines in patients with rheumatoid arthritis, proposed an algorithm for adjustment of immunomodulatory medications around the time of vaccination.

The lack of information on immune responses to SARS-CoV-2 vaccination in sarcoidosis indicates that studies to address this issue are urgently needed. The proposed investigation will begin to fill this critical knowledge gap by assessing both antibody and T cell responses to SARS-CoV-2 vaccination in individuals with sarcoidosis who are untreated and others who are treated with immunomodulatory agents in comparison to healthy control subjects.

Research Plan

General. Approval will be obtained from the Institutional Review Board of Northwestern University. The study will be registered with clinicaltrials.gov prior to the study start date.

Study Participants. Three groups of female and male subjects, all of whom will have completed primary vaccination, or primary vaccination plus booster vaccination, with one of the three SARS-CoV-2 vaccines currently authorized in the U.S. (BNT162b2 [Pfizer-BioNTech], mRNA-1273 [Moderna] or JNJ-78436735 [Johnson & Johnson]) at least 2 weeks previously, will be studied: 1) individuals with sarcoidosis not treated with immunosuppressive medications; 2) individuals with sarcoidosis treated with immunosuppressive medications, including systemic corticosteroids, methotrexate, azathioprine, mycophenolate mofetil, leflunomide, and anti-TNF monoclonal antibodies; and 3) individuals without sarcoidosis, other immune-mediated diseases, chronic lung disease, heart disease or malignancy, and not taking immunomodulatory medications [healthy controls]. Sarcoidosis subjects treated and not treated with immunosuppressive medications will recruited from established patients followed in the Pulmonary and Cardiology Clinics of the Northwestern Medicine Sarcoidosis Program. Healthy control subjects, matched for age and sex with the sarcoidosis subjects, will be recruited from members of the Northwestern Medicine community and the community at large. Demographic information, dates and type of SARS-CoV-2 vaccine received, and history of prior testing for SARS-CoV-2 infection or symptomatic COVID-19 will be recorded for all subjects. For sarcoidosis subjects, detailed information on method of sarcoidosis diagnosis, disease duration, past and present medical therapy for sarcoidosis, other current medications, co-morbid medical conditions, tobacco and other substance use, and occupation will be recorded. For healthy controls, current medications, past medical history, tobacco and other substance use, and occupation will likewise be recorded.

Specific Aim 1. Venous blood will be obtained from all subjects, and serum will separated, aliquoted and frozen for subsequent analysis. Serum anti-SARS-CoV-2 spike protein IgG will be measured following SARS-CoV-2 vaccination of individuals with sarcoidosis treated and not treated with immunosuppressive medications, and age- and sex-matched healthy controls using the LIAISON SARS-CoV-2 TrimericS IgG assay (Diasorin). This is a highly sensitive and specific second-generation assay for IgG antibodies to SARS-CoV-2 trimeric spike protein receptor binding domain. The assay has been calibrated against a separate SARS-CoV-2 virus neutralization assay, with a receiver operating characteristic area under the curve for detection of antibody with virus neutralization capacity of 0.996. The Diasorin TrimericS IgG assay received Emergency Use Authorization from the FDA on May 19.2021, and will replace the first-generation LIAISON SARS-CoV-2 S1/S2 IgG assay, which itself correlated most highly with virus neutralization capacity among five commercial SARS-CoV-2 antibody assays in a recent study. It should be noted that neutralizing antibody levels are highly predictive of immune protection from symptomatic SARS-CoV-2 infection. Serum samples will be stored frozen at -80°C and assayed as a batch when subject enrollment and sample acquisition are complete.

Power analysis: Extrapolating from data in a recent study of antibody responses to SARS-CoV2 vaccination in patients with rheumatic diseases on immunosuppressive therapies, the online sample size calculator ClinCalc.com was used to determine that up to 80 subjects per group will be required to detect a 20% reduction in average antibody level in either of the sarcoid groups compared to healthy controls, with a power of 0.80 at alpha 0.05.

Specific Aim 2. Peripheral blood mononuclear cells (PBMCs) will be isolated from anticoagulated venous blood of 10 subjects in each of the two sarcoidosis groups and healthy controls by Ficoll-Paque centrifugation, washed, resuspended in 10% dimethylsulfoxide/fetal bovine serum and cryopreserved at -80°C. SARS-CoV-2-specific CD4+ T cell activation will be assayed using PBMCs from sarcoidosis subjects treated and not treated with immunosuppressive medications, and age- and sex-matched healthy controls using the interferon-γ EliSpotPLUS assay (Mabtech). PBMCs will be stimulated with SARS-CoV-2 spike and nucleocapsid protein peptide pools (BEI Resources), or anti-cluster of differentiation 3 (CD3) antibody (Mabtech) as positive control, as described (19). PBMCs will remain cryopreserved at -80°C, then thawed, resuspended in culture medium, and assayed as a batch when subject enrollment and sample acquisition are complete. Alternatively, the T cell response to vaccination will be assessed in anticoagulated whole blood using the SARS-CoV-2 QuantiFERON assay (Qiagen).

Statistical Analysis. The significance of differences between group means will be determined by Analysis of Variance and Dunnett's Multiple Comparison Test. P < 0.05 will considered significant.

ELIGIBILITY:
Inclusion Criteria for Sarcoidosis Subjects:

* Age 18 years or older
* Diagnosis of sarcoidosis
* Receives clinical care at Northwestern Medicine in the Pulmonary Clinic, Cardiology Clinic or other Northwestern Medicine clinical unit
* Completed primary vaccination, or primary plus booster vaccination, with the Pfizer-BioNTech BNT162b2, Moderna mRNA-1273, or Johnson & Johnson JNJ-78436735 SARS-CoV-2 vaccine at least two weeks prior to enrollment

Exclusion Criteria for Sarcoidosis Subjects:

• Unable to provide informed consent in English

Inclusion Criteria for Healthy Controls:

* Age 18 years or older
* Completed primary vaccination, or primary plus booster vaccination, with the Pfizer-BioNTech BNT162b2, Moderna mRNA-1273, or Johnson & Johnson JNJ-78436735 SARS-CoV-2 vaccine at least two weeks prior to enrollment

Exclusion Criteria for Healthy Controls:

* Diagnosis of sarcoidosis or autoimmune diseases
* Diagnosis of chronic lung disease
* Diagnosis of heart disease
* Diagnosis of cancer
* Currently taking immunosuppressive medications
* Unable to provide informed consent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As above
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Humeral immune response | 2 weeks to 1 year following primary vaccination, or primary + booster vaccination
  Anti-spike IgG level
Cell-mediated immune response | 2 weeks to 1 year following primary vaccination, or primary + booster vaccination
  Level of interferon-gamma release by peripheral blood T cells in response to SARS-CoV-2 peptide stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sporn, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simon D, Tascilar K, Fagni F, Kronke G, Kleyer A, Meder C, Atreya R, Leppkes M, Kremer AE, Ramming A, Pachowsky ML, Schuch F, Ronneberger M, Kleinert S, Hueber AJ, Manger K, Manger B, Berking C, Sticherling M, Neurath MF, Schett G. SARS-CoV-2 vaccination responses in untreated, conventionally treated and anticytokine-treated patients with immune-mediated inflammatory diseases. Ann Rheum Dis. 2021 Oct;80(10):1312-1316. doi: 10.1136/annrheumdis-2021-220461. Epub 2021 May 6. PMID 33958324